CLINICAL TRIAL: NCT01895478
Title: Adaptation of the Pediatric Asthma Control & Communication Instrument (PACCI) in a Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Aris Garro, Pediatric Emergency Medicine Attending Physician, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 210394
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
Keywords: asthma; pediatrics; control; medication adherence
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PACCI-ED (Experimental): PACCI-ED attendings were given the PACCI-ED use intervention.
  Interventions: Behavioral: PACCI-ED use
- Control (No Intervention): Control attendings were not given the PACCI-ED use intervention.

INTERVENTIONS:
Behavioral: PACCI-ED use — Attending physicians were allowed to view the patient's PACCI-ED prior to completing the assessment form. Attendings were told at the time of the child's ED visit that the PACCI-ED is used to assess a child's asthma control and medication adherence, and that they could use it to complete the outcomes assessment form.
  Arms: PACCI-ED

SUMMARY:
This study examined whether the Pediatric Asthma Control and Communication Instrument for the Emergency Department (PACCI-ED), a 12-item questionnaire, can help doctors in the emergency department accurately assess a child's asthma control.

This study involved an intervention with the doctors in the emergency department of an urban pediatric hospital. The intervention was done when one of the doctors involved in the study treated a child aged 1-17 years for an asthma exacerbation. Parents answered questions on the PACCI-ED about their children's asthma. Half of the doctors were allowed to see the PACCI-ED results and half were not. The two groups of doctors were compared on their ability to correctly identify asthma control categories, whether a child's asthma was worsening or improving, whether the family was administering controller medications as often as they should, and how much burden the child's asthma was for the family.

ELIGIBILITY:
Inclusion Criteria:

* Child presented to study institution emergency department during study period
* Child was 1 - 17 years-old
* Child has physician-diagnosed asthma by parent report
* Attending physician for child believed emergency department visit was due to asthma
* Attending physician for child completed informed consent and was randomized to PACCI-ED or control group at beginning of study

Exclusion Criteria:

* Child has major pulmonary or cardiac co-morbid illness
* Family of child was non-English speaking
* Child was triaged to the med-trauma bay for severe respiratory distress

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Asthma Control | 1 day (Assessment occurs at a single time during emergency department visit)
  Attending physician answered "Which of the following best describes this patient's asthma control over the past 12 months?" (RESPONSES: Controlled, partly controlled, mildly uncontrolled, moderately uncontrolled, severely uncontrolled). Responses were compared to equivalent categories of control based on PACCI algorithm.

SECONDARY OUTCOMES:
Asthma Trajectory | 1 day (Assessment occurs at a single time during emergency department visit)
  Attending physician answered "Which of the following best describes the changes in this patient's asthma status over the past 12 months?" (RESPONSES: No change, getting worse, getting better). Responses were compared to equivalent categories of trajectory based on PACCI algorithm.
Medication Adherence | 1 day (Assessment occurs at a single time during emergency department visit)
  Attending physician answered "In your clinical judgment, during the past week, how often does this patient use his/her daily controller asthma medicine?" (RESPONSES: Not at all (0 days/week), sometimes (1-3 days/week), most of the time (4-6 days/week), all of the time (7 days/week)). Responses were compared to equivalent categories of medication adherence based on PACCI algorithm.
Asthma burden to family | 1 day (Assessment occurs at a single time during emergency department visit)
  Attending physician answered "Which of the following best describes how burdensome to the caregiver this patient's asthma has been over the past 12 months?" (RESPONSES: Not at all burdensome, somewhat burdensome, very burdensome). Responses were compared to equivalent categories of asthma burden based on PACCI algorithm.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital / Hasbro Children's Hospital, Providence, Rhode Island, United States